CLINICAL TRIAL: NCT04751227
Title: Modafinil for Wakefulness in the Critical Care Units and COVID-19 Patients at a Tertiary Care Saudi Hospital
Brief Title: Modafinil for Wakefulness in the Critical Care Units
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, MARWA RIDHA AMER, ICU clinical Pharmacist, Adjunct Assistance professor- college of medicine Alfaisal university, King Faisal Specialist Hospital & Research Center
Other Study IDs: RAC # 2201230
Record Dates: First submitted 2021-02-04; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Critical Illness; COVID-19; Cognitive Dysfunction
MeSH Terms: conditions — Critical Illness; COVID-19; Cognitive Dysfunction | interventions — Modafinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: Modafinil 100-200 mg daily for wakefulness in a cohort of adult patients admitted to our COVID and non-COVID intensive care unit (ICU) between January 2017 and June 2020
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — 100-200 mg oral daily for for Wakefulness in the Critical Care Units

SUMMARY:
It has been well documented that patients in the intensive care unit (ICU) are susceptible to developing neurocognitive and musculoskeletal complications because of various factors, including the nature of the critical illness, medications, over-sedation, and pain. Neuro-stimulants are used to speed up physical and mental processes through the increase in neurotransmitter, which translates into increase in arousal, wakefulness, attention, memory, mental and motor processing speed. The investigators reviewed the literature and described the clinical characteristics for a case series of adult patients admitted to COVID and non-COVID ICU between January 2017 and June 2020, who received modafinil to promote wakefulness and improve cognition at the King Faisal Specialist Hospital and Research Centre (KFSH&RC) in Riyadh, Saudi Arabia. The secondary goals to describe the change of Glasgow Coma Scale (GCS) before and after the start of modafinil therapy, ICU and hospital length of stay, discharge disposition, adverse drug effects, and mortality rate.

ELIGIBILITY:
Inclusion Criteria:

1. ICU patients 18 years and older
2. admitted to COVID and non-COVID units between January 2017 and June 2020
3. ICU stay for at least 48 hours
4. started on modafinil during ICU stay for at least 48 h
5. required ventilatory support.

Exclusion Criteria:

* Those who did not receive modafinil or received modafinil for indications other than ICU wakefulness

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID ICU and non-COVID ICU units (medical, surgical, transplant/oncology ICUs).
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-11-22 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Median change in of Glasgow Coma Scale (GCS) | 48 hours before modafinil therapy and 7 days after modafinil therapy
  Describe the median change in Glasgow Coma Scale (GCS) before and after modafinil therapy. The GCS is used to assess and communicate changes in mental status and to measure the duration of coma. The Glasgow Coma Scale is comprised of the individual components, e.g. "eye(4) verbal(5) motor (6)". Glasgow Coma Score is calculated by addition of the total points selected under each component (eye, verbal, motor) score can range from 1 and 15

SECONDARY OUTCOMES:
adverse drug reactions (ADRs) | until ICU discharge, 90 days or death whichever occurs first.
  Number of patients started on antipsychotics and with possible adverse drug reactions (ADRs) related to modafinil including nervousness, agitation, delirium, hypersensitivity, and drug rash. Naranjo scale was used to evaluate the causality of ADRs and modafinil therapy
Duration of Mechanical Ventilation | From Intubation to extubation date and off Mechanical Ventilation or until ICU discharge, death, or 90 days whichever occurs first. ]
  To assess whether modafinil can help to shorten the time of being in breathing tube and ventilator (duration of mechanical ventilation )
ICU Length of stay (LOS) | until ICU discharge, 90 days or death whichever occurs first.
  To describe ICU LOS
Hospital Length of Stay (LOS) | until hospital discharge, 90 days or death whichever occurs first.
  To describe hospital LOS
Mortality rate | 28 days and 90 days
  Death that occurs during 28 days and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Marwa R Amer, PharmD, BCPS,BCCCP, Principal Investigator — KFSHRC
Locations (1):
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia